CLINICAL TRIAL: NCT05454059
Title: Investigation of Salivary Ceramide-1-Phosphate and Prostaglandin E2 Levels in Periodontitis Patients With Poorly and Well-Controlled Type 2 Diabetes and Effect of Non-Surgical Periodontal Treatment: A Randomized Controlled Clinical Trial
Brief Title: Salivary C1P and PGE2 Levels in Periodontitis Patients With T2DM and Effect of Non-Surgical Periodontal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, SELMAN YILMAZ CICEK, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/598
Record Dates: First submitted 2022-07-01; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Periodontitis; Type 2 Diabetes
Keywords: saliva; prostaglandin e2; ceramide-1-phosphate; non-surgical periodontal treatment; phase I periodontal therapy; saliva biomarker; metabolic control; HbA1c; PGE2; C1P; periodontitis; type 2 diabetes mellitus
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2 | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Intervention Model Description: A total of 102 (n=102) individuals were included in the study and were divided into 6 groups. The control groups of our study were Group 1 (HH), which included 17 both systemically healthy and periodontally healthy normoglycemic individuals, Group 2 (HP), which included 17 systemic healthy with Grade A periodontitis. Periodontally healthy T2DM patients were divided into two groups according to their HbA1c levels, and 17 patients with HbA1c levels below 7% were grouped as Group 3 (T2D+H), and 17 patients with HbA1c above 7% and 7% were grouped as Group 5 (T2D-H). 17 patients with T2DM with Grade B periodontitis with an HbA1c below 7% in the last three months were included in Group 4 (T2D+P), and 17 patients T2DM and periodontitis with an HbA1C value above 7% were included in Group 6 (T2D-P).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group 1 (HH) (Active Comparator): 17 systemically healthy + periodontally healthy (normoglycemic)
  Interventions: Diagnostic Test: ELISA Test; Other: Periodontal Examination; Other: Saliva Sample Collection
- Group 2 (HP) (Experimental): 17 systemic healthy + grade A periodontitis
  Interventions: Procedure: Non-surgical periodontal treatment; Diagnostic Test: ELISA Test; Other: Periodontal Examination; Other: Saliva Sample Collection
- Group 3 (T2D+H) (Active Comparator): 17 T2DM (HbA1c<%7) + periodontally healthy
  Interventions: Diagnostic Test: ELISA Test; Other: Periodontal Examination; Other: Saliva Sample Collection; Diagnostic Test: HbA1c Level
- Group 4 (T2D+P) (Experimental): 17 T2DM (HbA1c<%7) + grade B periodontitis
  Interventions: Procedure: Non-surgical periodontal treatment; Diagnostic Test: ELISA Test; Other: Periodontal Examination; Other: Saliva Sample Collection; Diagnostic Test: HbA1c Level
- Group 5 (T2D-H) (Active Comparator): 17 T2DM (HbA1c≥%7) + periodontally healthy
  Interventions: Diagnostic Test: ELISA Test; Other: Periodontal Examination; Other: Saliva Sample Collection; Diagnostic Test: HbA1c Level
- Group 6 (T2D-P) (Experimental): 17 T2DM (HbA1c≥%7) + grade C periodontitis
  Interventions: Procedure: Non-surgical periodontal treatment; Diagnostic Test: ELISA Test; Other: Periodontal Examination; Other: Saliva Sample Collection; Diagnostic Test: HbA1c Level

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Routine non-surgical periodontal treatment will be applied to patients with periodontitis. The main aim of non-surgical periodontal treatment is to protect, heal and maintain the existing dentition. For this purpose, using manual, sonic or ultrasonic instruments, microbial dental plaque and calculus are removed by tooth surface cleaning and root surface straightening.
  Other Names: phase I periodontal therapy; scaling and root planing; full mouth debridement
  Arms: Group 2 (HP); Group 4 (T2D+P); Group 6 (T2D-P)
Diagnostic Test: ELISA Test — C1P and PGE2 levels in saliva samples obtained, and will be examined by ELISA test.
Other: Periodontal Examination — All diagnostic procedures were performed with examination instruments (periodontal probe, dental mirror, x-ray device, etc.). Periodontal clinical index measurements (PI, GI, BOP, PPD, CAL) recorded from all teeth. Routine panoramic radiographs were taken from all patients to determine alveolar bone resorption. Vertical/horizontal bone losses on the radiographs were evaluated and used in the diagnosis of periodontitis.
Other: Saliva Sample Collection — Saliva samples were collected from all subjects in the morning. Unstimulated saliva from each patient was collected by standard defined spitting method without stimulation.
Diagnostic Test: HbA1c Level — Measurement of HbA1c levels from blood tests
  Arms: Group 3 (T2D+H); Group 4 (T2D+P); Group 5 (T2D-H); Group 6 (T2D-P)

SUMMARY:
Diabetes and periodontal disease are the most common chronic multifactorial and inflammatory diseases in humans, and there is a bidirectional relationship between type 2 diabetes and periodontitis. With the negative effects of the control of these two diseases, it results in an increase in the severity of diabetes and periodontitis, and they affect many systems together. To elucidate the role of ceramide, which is one of the possible biochemical mechanisms between diabetes and the degree of glycemic control and periodontitis, in inflammation. Aim of this study is the measurement of C1P and PGE2 in saliva and the effect of non-surgical periodontal treatment, which includes the degree of control of diabetes, oral hygiene education, tooth surface cleaning and root surface arrangement, on 3 months.

A total of 102 subjects were included. Clinical periodontal measurements, saliva samples were collected from each individual at baseline and 3 months after non-surgical periodontal treatmet in periodontitis groups. Salivary C1P and PGE2 levels were determined by enzyme-linked immunosorbent assay (ELISA) method.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 30-65
* Have not received periodontal treatment in the last 6 months,
* Does not have any systemic disease and does not use drugs,
* Not using local or systemic antibiotics in the last 3 months,
* HbA1c <%7 for the controlled T2DM group,
* HbA1c ≥7% for the uncontrolled T2DM group,
* For female patients who are not in the pregnancy or lactation period,
* Non-smoker,
* Not regularly using mouthwash/mouthwash.

Exclusion Criteria:

* Not being willing to participate in the study,
* Under 30 years old, over 65 years old
* Having any systemic disease affecting the periodontal condition,
* To use any medication that may affect the inflammatory process in the last 3 months,
* Using local or systemic antibiotics in the last 3 months,
* To have had periodontal treatment in the last 6 months,
* Being in pregnancy or lactation period for female patients,
* Using mouthwash regularly
* Smoking

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
PGE2 levels in saliva | baseline to 3 months after treatment
  Change in saliva PGE2 levels from baseline to 3 months after non-surgical periodontal treatment
C1P levels in saliva | baseline to 3 months after treatment
  Change in saliva C1P levels from baseline to 3 months after non-surgical periodontal treatment
HbA1c levels | baseline to 3 months after treatment
  Blood test in routine biochemistry laboratory for evaluation of the change in HbA1c levels of patients with type 2 diabetes from baseline to 3 months after non-surgical periodontal treatment

SECONDARY OUTCOMES:
Plaque index (PI) | baseline to 3 months after treatment
  The changes in PI from baseline to 3 months after non-surgical periodontal treatment
Bleeding on probing index (BOP) | baseline to 3 months after treatment
  The changes in BOP from baseline to 3 months after non-surgical periodontal treatment
Gingival index (GI) | baseline to 3 months after treatment
  The changes in GI from baseline to 3 months after non-surgical periodontal treatment
Probing pocket depth | baseline to 3 months after treatment
  The changes in probing pocket depth from baseline to 3 months after non-surgical periodontal treatment
Clinical attachment level (CAL) | baseline to 3 months after treatment
  The changes in CAL from baseline to 3 months after non-surgical periodontal treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No